CLINICAL TRIAL: NCT05844241
Title: The Effect of Auditory Interventions on Anxiety and Agitation in People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucid, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LUC101A
Record Dates: First submitted 2023-04-10; First posted 2023-05-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-05

CONDITIONS: Mild to Moderate Dementia
MeSH Terms: interventions — Sound Recordings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music and Theta Auditory Beat Stimulation (ABS) (Experimental): Participants listen to 30 minutes of personalized music with theta auditory beat stimulation (ABS).
  Interventions: Other: Music and Theta Auditory Beat Stimulation
- Audiobooks (Active Comparator): Participants listen to a 30-minute audiobook.
  Interventions: Other: Audiobooks

INTERVENTIONS:
Other: Music and Theta Auditory Beat Stimulation — Listening to music and ABS for 30 minutes.
  Arms: Music and Theta Auditory Beat Stimulation (ABS)
Other: Audiobooks — Listening to audiobooks for 30 minutes
  Arms: Audiobooks

SUMMARY:
The greying of the world is leading to a rapid acceleration in both the healthcare costs and caregiver burden that are associated with dementia. There is an urgent need to develop new, easily scalable modalities of support to reduce agitation and anxiety in those with dementia. There is evidence that music interventions reduce agitation and anxiety in those with dementia. LUCID has developed a novel digital music therapeutic product that uses a reinforcement learning AI agent to curate and personalize the musical playlist while incorporating binaural theta auditory beat stimulation (ABS) to reduce anxiety and agitation in those with dementia. This study will be conducted remotely with study hardware (tablets and Bluetooth speakers) being shipped to caregivers/participants' homes. The study will take place over a 2-week period, with participants completing 4 one-hour sessions per week along with an additional 1-hour follow-up interview session. Forty-eight participants with mild to moderate dementia (as defined by the Montreal Cognitive Assessment) will be evenly randomized to one of two conditions. The control condition consists of a selection of 30-minute audiobooks which the participant has the freedom to select from. The experimental condition consists of music and binaural ABS curated by LUCID's AI system. Participants' caregivers will complete baseline questionnaires assessing the participants' anxiety, agitation, and mood. They will also complete these questionnaires before and after each experimental session. The investigators hypothesize that the LUCID AI music curation system will have a greater agitation and anxiety reduction compared to the audiobook control condition.

DETAILED DESCRIPTION:
The greying of the world is leading to a rapid acceleration in both the healthcare costs and caregiver burden that are associated with dementia. There is an urgent need to develop new, easily scalable modalities of support to reduce agitation and anxiety in those with dementia. There is evidence that music interventions reduce agitation and anxiety in those with dementia. LUCID has developed a novel digital music therapeutic product that uses a reinforcement learning AI agent to curate and personalize the musical playlist while incorporating binaural theta auditory beat stimulation (ABS) to reduce anxiety and agitation in those with dementia. This study will be conducted remotely with study hardware (tablets and Bluetooth speakers) being shipped to caregivers/participants' homes. The study will take place over a 2-week period, with participants completing 4 one-hour sessions per week along with an additional 1-hour follow-up interview session. Forty-eight participants with mild to moderate dementia (as defined by the Montreal Cognitive Assessment) will be evenly randomized to one of two conditions. The control condition consists of a selection of 30-minute audiobooks which the participant has the freedom to select from. The experimental condition consists of music and binaural ABS curated by LUCID's AI system. Participants' caregivers will complete baseline questionnaires assessing the participants' anxiety, agitation, and mood. They will also complete these questionnaires before and after each experimental session. Participants and their caregivers will schedule a Zoom call with a Research Assistant (RA) to assist them during their first onboarding session and go over study expectations and participants' rights. Participants/caregivers have access to and the ability to communicate and schedule meetings with RAs at any time should any issues arise over the course of the study. The investigators hypothesize that the LUCID AI music curation system will have a greater agitation and anxiety reduction compared to the audiobook control condition.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate Dementia (mild: Montreal Cognitive Assessment (MOCA) scores (18-25); moderate: MOCA scores (10-17)))

Exclusion Criteria:

* Unmanaged hearing loss (defined as average pure-tone average threshold of 35 dB HL or greater without the use of hearing instruments or personal sound amplification product)
* Severe Tinnitus
* Hyperacusis

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Cohen Mansfield Agitation Index | 2 weeks
  The purpose of this scale is to assess the frequency of manifestations of agitated behaviors in elderly persons. Minimum score: 14, Maximum score: 70. Higher score indicates a worse outcome (increased agitation).

SECONDARY OUTCOMES:
Rating of Anxiety in Dementia | 2 weeks
  A rating scale to measure anxiety in those that suffer from dementia. Minimum value: 0, Maximum value: 54. Higher score indicates worse outcome (increased anxiety)
Cornell Brown Scale for Quality of Life in Dementia | 2 weeks
  A scale that measures the quality of life of dementia patients. Minimum score: -38. Maximum score: 38. Higher score indicates better outcome (increased quality of life)
Zarit Caregiver Burden Interview | 2 weeks
  A scale that measures the caregiver burden of those that care for people with dementia and other ailments. Minimum score: 0, Maximum score: 88, Higher score indicates a worse outcome (higher caregiver burden).
Positive and Negative Affect Scale | 30 minutes
  The positive and negative affect scale is a good measure of a person's current mood. This scale generates two scores: 1) Positive affect (a higher score indicates a better outcome), scores range from 10-50. 2) Negative affect (higher score indicates worse outcome), scores range from 10-50.
Overt Agitation Severity Scale | 30 minutes
  A scale that identifies and measures the severity of agitated behavior in those with dementia/Alzheimer's disease. Minimum score: 0, Maximum score: 48. Higher score indicates a worse outcome (higher agitation symptoms).
Digit Span Forward | 30 minutes
  A cognitive measure of working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Adiel Mallik, PhD, Principal Investigator — Lucid, Inc.
Locations (1):
- LUCID Therapeutics, Toronto, Ontario, Canada